CLINICAL TRIAL: NCT04145102
Title: Evaluation of the Remineralizing and Antibacterial Effect of Natural Versus Synthetic Materials on Deep Carious Dentin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Dalia Mohamed Elasser, Doaa Elsharkawy,Assistant Professor of operative department, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC18-076
Record Dates: First submitted 2019-10-19; First posted 2019-10-30 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Dentin Caries
Keywords: remineralization; carious dentin; natural products; antibacterial effect
MeSH Terms: conditions — Dental Caries | interventions — Propolis; silver diamine fluoride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- negative control (No Intervention): restoration will applied without any treatment
- hesperidine (Experimental): hesperidine will be applied for remaining caries then restoration will be applied
  Interventions: Other: hesperidine
- propolis (Experimental): propolis will be applied for remaining caries then restoration will be applied
  Interventions: Other: propolis
- silver diamine fluoride (Experimental): silver diamine fluoride will be applied for remaining caries then restoration will be applied
  Interventions: Other: silver diamine fluoride

INTERVENTIONS:
Other: hesperidine — used for antibacterial and reminerlization assesment
  Arms: hesperidine
Other: propolis — used for antibacterial and reminerlization assesment
  Arms: propolis
Other: silver diamine fluoride — used for antibacterial and reminerlization assesment
  Other Names: riva star
  Arms: silver diamine fluoride

SUMMARY:
The present study will be performed to evaluate:

1. The remineralizing effect of natural materials versus synthetic materials on deep carious dentin after selective caries removal.
2. The antibacterial effect of natural materials versus synthetic materials on deep carious dentin.

DETAILED DESCRIPTION:
This study will be conducted on 64 teeth selected from patients according to inclusion and exclusion criteria. They will be selected from the dental clinic in faculty of dental medicine, Al-Azhar University. The procedure will be explained and written informed consent will be obtained from each patient. The possible discomforts, risks, and benefits will be fully explained to the patients. Ethical committee approval will be obtained.

Protocol of caries removal will be removed Subsequently, the central cariogenic biomasses and superficial part of the necrotic and demineralized dentin will be then excavated, leaving the last carious affected dentin layer.

Sample grouping:

The patients will be randomly assigned into four main groups according to the material used (16 for each) then each group will be subdivided into two subgroups (n=8) according to time of treatment (B1) after one month,(B2) after three month.

A1: cavities will be treated by propolis extract then sealed directly by temporary conventional glass ionomer.

A2: cavities will be treated by hesperidin then sealed directly by temporary conventional glass ionomer.

A3: cavities will be treated with Silver diamine fluoride then sealed directly by temporary conventional glass ionomer.

A4: cavities will be sealed directly by temporary restorative material (conventional glass ionomer) without any treatment.

Evaluation of the microbiological effect Dentine samples will be collected from the base of the cavity using sterile spoon excavator from the four groups for baseline bacteriological assessment immediately after excavation, then another sample will be taken after one month for each subgroup (B1)and three months of treatment for each subgroup (B2).

Evaluation of the remineralization effect Each group will be assessed radiographically immediately at base line (B0), after one month (B1) and three months (B2) to evaluate the dentin remineralization.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have active deep carious lesion.
* clinical and radiographic examinations of carious lesions.

Exclusion Criteria:

* Teeth with pulpal involvement
* Teeth with abscess
* Teeth with pain or swelling
* Teeth with developmental disorders
* Teeth with adjacent soft tissue lesions
* patients with systemic illness will be excluded

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Remineralizing and Antibacterial Effect of Natural Versus Synthetic Materials on Deep Carious Dentin | antibacterial and reminerlizing effect will be evaluated after three monthes
  antibacterial effect will be evaluated by bacterial count at base line and after three months reminerliazation effect will be evaluated by radiographes

CONTACTS AND LOCATIONS:
Locations (1):
- Alazher university, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anani H, Elasser D, Niazy M, Jamil W, Elsharkawy D. Evaluation of the remineralization and antibacterial effect of natural versus synthetic materials on deep carious dentin: A randomized controlled trial. Dent Med Probl. 2023 Jan-Mar;60(1):87-97. doi: 10.17219/dmp/147075. PMID 37023336